CLINICAL TRIAL: NCT06157476
Title: Stretch-shortening Cycle Exercise: a Clinical Trial Investigating Its Role for Strength, Bone Mineral Density, and Functional Capacity in Children With Obstetric Brachial Plexus Injury
Brief Title: Stretch-Shortening Cycle Exercise: Potential Implications For Children With Obstetric Brachial Plexus Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0021/0015
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Erb Palsy
MeSH Terms: conditions — Brachial Plexus Neuropathies | interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: A prospective, two-arm, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind protocol. The researcher who collected the data was blind to the allocation of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSC-Ex group (Experimental): Children in this group received the SSC-Ex program
  Interventions: Other: Stretch-shortening exercise
- Control group (Active Comparator): Children in this group received the standard exercise program.
  Interventions: Other: Standard exercise program

INTERVENTIONS:
Other: Stretch-shortening exercise — The SSC-Ex program was conducted for 35 minutes/session twice weekly over 12 weeks. The program was directed by a pediatric physical therapist in accordance with the safety performance guidelines defined by the American Academy of Pediatrics and the US National Strength and Conditioning Association. The program consisted of ten unilateral and bilateral upper extremity exercises in the form of push-ups and ball slams/throws/passes activities and was preceded by a warm-up for 5 minutes and ended with a cool-down for 5 minutes.
  Arms: SSC-Ex group
Other: Standard exercise program — The standard exercise program lasted for 35 minutes/session and repeated two times a week for 12 consecutive weeks. The program was conducted by a pediatric physical therapist and consisted of flexibility exercises, strength training, weight-bearing exercises, proprioceptive neuromuscular facilitation, manual guidance, and functional training.
  Arms: Control group

SUMMARY:
This study was set out to evaluate the effect of a 12-week stretch-shortening cycle exercise (SSC-Ex) on muscle strength, bone mineral density, and upper extremity function in children with obstetric brachial plexus injury (OBPI). Fifty-six patients with OBPI were randomly allocated to the SSC-Ex group (n = 28, received SSC-Ex program, twice/week, over 12 weeks) or the control group (n = 28, received standard exercise program). Both groups were assessed for muscle strength, bone health, and upper extremity function before and after treatment.

DETAILED DESCRIPTION:
Fifty-six children with OBPI were recruited from the Physical Therapy Outpatient Clinic of Prince Sattam Bin Abdulaziz University and three referral hospitals in Riyadh provenience, Saudi Arabia. The study included children who had a confirmed diagnosis of upper arm type of OBPI, classified as level I or II per Narakas classiﬁcation system, aged 10-16 years, had a functional level of grade III according to the Mallet scoring system, and were consuming a balanced diet. Children who had a history of corrective neuromotor or musculoskeletal surgery, shoulder dislocation/subluxation, calcium supplements, or cognitive issues were excluded.

Outcome measures

1. Muscle strength: The peak isometric muscle strength of the shoulder flexors, abductors, external rotators, elbow flexors, and extensors was measured using a hand-held dynamometer.
2. Bone mineral properties: Bone mineral density and bone mineral content of the humeral, radial, and ulnar shafts were measured through Dual-Energy X-ray Absorptiometry (DEXA) scanning.
3. Upper-extremity function: The functional performance was assessed using the brachial plexus outcome measure (BPOM) activity scale.

The SSC-Ex group received a 12-week therapist-led SSC-Ex training, for approximately 35 minutes per session, two times a week for 12 consecutive weeks, in conformity with the National Strength and Conditioning Association guidelines and American Academy of Pediatrics safety standards. The SSC-Ex program consisted of ten unilateral and bilateral upper extremity exercises in the form of push-ups and ball slams/throws/passes activities. The SSC-Ex program preceded with a warm-up for 5 minutes and ended with a cool-down for 5 minutes. The control group received the standard exercise program, 35 minutes per session, two times a week for 12 consecutive weeks. The program consisted of flexibility exercises, strength training, weight-bearing exercises, proprioceptive neuromuscular facilitation, manual guidance, and functional training.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of upper arm type of OBPI.
* Narakas classiﬁcation level I or II.
* Functional level of grade III per the Mallet scoring system.
* Age between 10-16 years.

Exclusion Criteria:

* History of neuromotor or musculoskeletal surgery.
* Shoulder subluxation/dislocation.
* Past fracture involving the upper extremities.
* Calcium supplement intake.
* Inability to adhere to the scheduled program.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2021-03-14 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 2 months
  The peak isometric muscle strength (Kg) was measured using a hand-held dynamometer.
Bone mineral density | 2 months
  The amount of bone mineral divided by the bone scanned area (gm/cm2). It was assessed within the humeral, radial, and ulnar shafts using DEXA scanning.
Bone mineral content | 2 months
  It is the amount of bone mineral in bone tissue (g/cm). It was calculated by summing the bone mineral density values over the projected area. It was also measured within the humeral, radial, and ulnar shafts using DEXA scanning.

SECONDARY OUTCOMES:
Functional performance | 2 months
  The affected arm functionality was assessed using the brachial plexus outcome measure. activity scale [an 11-item performance-based measure with five-point ordinal ratings for each item (I = cannot complete the task and 5 = complete the activity with normal pattern); higher scores denote better performance, with 55 being the maximum attainable score].

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K. Elnaggar, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No